CLINICAL TRIAL: NCT02667691
Title: Evaluation of SODB®, Associated With a Caloric Restriction, in Metabolic Adaptations in Overweight Women: Randomized Double-blind Study Versus Placebo
Brief Title: Evaluation of SODB® in Metabolic Adaptations in Overweight Women
Acronym: SORESCAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bionov (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2014-A01974-43
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Overweight
Keywords: superoxyde dismutase; melon concentrate; oxydative stress; overweight women
MeSH Terms: conditions — Overweight | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SODB Dimpless-caloric restriction (Experimental): This arm receives daily two capsules of SODB Dimpless 40mg containing 480 UI of superoxide dismutase (SOD), associated with a moderate caloric restriction.
  Interventions: Dietary Supplement: SODB Dimpless; Other: caloric restriction
- Placebo-caloric restriction (Placebo Comparator): This arm receives daily two capsules Placebo containing excipients only, associated with a moderate caloric restriction.
  Interventions: Dietary Supplement: Placebo; Other: caloric restriction

INTERVENTIONS:
Dietary Supplement: SODB Dimpless — Subjects are supplemented with SODB, daily over 3 Months. Each volunteer was seen for the 4 visits: - visit of pre-inclusion, - visit V1, so-called inclusion visit, - visit V2 at 1,5 months and - visit V3 at 3 months
  Arms: SODB Dimpless-caloric restriction
Dietary Supplement: Placebo — Subjects are supplemented with placebo, daily over 3 Months. Each volunteer was seen for the 4 visits: - visit of pre-inclusion, - visit V1, so-called inclusion visit, - visit V2 at 1,5 months and - visit V3 at 3 months
  Arms: Placebo-caloric restriction
Other: caloric restriction — Caloric recommendation reduced by 20%

SUMMARY:
The objective of this study is to evaluate the influence of a 3 months SODB® supplementation in adipose tissue modulations of overweight women, in comparison to a placebo.

DETAILED DESCRIPTION:
Beneficial experimental results have already been obtained with SODB®. That is why, the investigators expect several effects of SODB® here. Indeed, this clinical study could show that SODB® is able to induce endogenous antioxidant defence, and then reduce oxidative stress generally observed in overweight adipose tissue.

Moreover, this study could evaluate the impact of a decrease in oxidative stress on the others overweight-induced disorders, such as insulin resistance, inflammation, fibrosis, lipolyse alterations.

ELIGIBILITY:
Inclusion Criteria:

* overweight women (IMC 25-30 kg/m2)
* stable weight (variation <5% over the last 3 months)
* age between 25 and 50 years old
* cellulite grade ≥ 2
* women with genital activity
* regular menstrual cycles (28 ± 2 days over the last 3 months)
* women with efficient contraception (oral, intra-uterine, ligature trunks or other surgery) - same contraception over the last 3 months
* women having given her free, informed and express consent.
* affiliated with a social security insurance or beneficiary of such an insurance system.
* glycemia < 1,26g/l
* Arterial blood pression < 140/90 mm Hg or stable for at least 2 months
* LDL cholesterol <1,90g/l
* triglycerides <2,50g/l

Exclusion Criteria:

* untreated dyslipidemia
* unstable hypertension
* type 1 or 2 diabetes
* any history of bariatric surgery
* any history of unstable thyroidian diseases
* any troubles of hemostasis
* any allergy to utilized antiseptic, xylocaine, or to one of the compounds of the experimental or placebo product
* excessive coffee consumption (> 6 cups/day)
* consumption of drinks containing xanthic bases (> 0.5 l/day)
* consumption of drinks containing grapefruit juice (> 0.5 l/day)
* consumption of drinks containing plants (> 2 l/day)
* medication with draining, lipolytic, anorexigenic activity
* current or recent (in the previous month) antioxidant supplementation (vitamine A, C, E, beta-carotene, lutein, lycopene, selenium)
* recent (in the previous year) local anti-cellulite treatment
* thigh liposuction in the last 2 years
* under current anticoagulant treatment
* under current neuroleptic treatment
* under current corticotherapy (local or systemic) treatment
* under current diuretic treatment
* under current antiinflammatory treatment that cannot be interrupted
* under current treatment which interferes with autonomous nervous system and lipids metabolism
* triglycérides > 2.50g/l
* LDL cholesterol >1.90
* positive serology for hepatitis B, C and HIV
* consumption of more than 66g/day of alcohol
* venous fragility not allowing to support catheters during the visits.
* adult protected by the law
* any subject who participated to a clinical assay within the 3 months.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline adipocytes size at 3 months | Evaluation performed at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by immunohistology in subcutaneous abdominal adipose tissue.

SECONDARY OUTCOMES:
Evaluation of body composition | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by Dual energy X-ray absorptiometry (DEXA).
Evaluation of cellulite grade | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by a score.
Evaluation of body weight | Evaluation at inclusion day (V1), after 1.5 months of treatment (V2), and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by body weight measurements.
Evaluation of glycemia | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by glucose measurements.
Evaluation of insulinemia | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by insulin measurements.
Evaluation of non esterified fatty acids level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by non esterified fatty acids measurements.
Evaluation of triglycerides level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by triglycerides measurements.
Evaluation of cholesterol level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by cholesterol measurements.
Evaluation of glycerol level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by glycerol measurements.
Evaluation of adipokines level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by adipokines measurements.
Evaluation of C-reactive protein (CRP) level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by CRP measurements.
Evaluation of albumin level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by albumin measurements.
Evaluation of prealbumin level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by prealbumin measurements.
Evaluation of retinol binding protein (RBP) level | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by RBP measurements.
Evaluation of adipocytes size | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by immunohistology in subcutaneous gluteo-femoral adipose tissue.
Evaluation of adipocytes number | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by immunohistology in subcutaneous abdominal and gluteo-femoral adipose tissues.
Evaluation of fibrosis | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by immunohIstology (red sirius coloration) in subcutaneous abdominal and gluteo-femoral adipose tissues.
Evaluation of macrophage infiltration | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by immunohistology in subcutaneous abdominal and gluteo-femoral adipose tissues.
Adipose tissue secretions of glycerol | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by glycerol measurements in subcutaneous abdominal adipose tissue
Adipose tissue secretions of non esterified fatty acids | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by non esterified fatty acids measurements in subcutaneous abdominal adipose tissue
Adipose tissue secretions of adipokines | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation performed by adipokines measurements in subcutaneous abdominal adipose tissue
Adipose tissue genetic profile modifications | Evaluation at inclusion day (V1) and after 3 months of treatment at the end of the study (V3).
  Evaluation of genes (all human known genes tested) differentially expressed in the two arms of subjects performed by DNA microarrays in subcutaneous abdominal adipose tissue.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events | Evaluation at inclusion day (V1), after 1.5 months of treatment (V2), and after 3 months of treatment at the end of the study (V3).
  All the adverse events occured throughout the study analyzed in order to know the number of participants only with treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thalamas, Principal Investigator — CIC Hopital Purpan

IPD SHARING:
Plan to Share IPD: Undecided